CLINICAL TRIAL: NCT05452304
Title: A Phase 1 Randomised, Double-Blind, Placebo-Controlled 3 Part Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7798 Following Single Ascending Dose Administration and Repeat Dose Administration in Healthy Subjects (Including Japanese and Chinese Subjects), and Patients With Crohn's Disease
Brief Title: AZD7798 Safety, Tolerability, and Pharmacokinetics After a Single Ascending and Repeat Dose Administrations to Healthy Subjects, and Patients With Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9690C00001; 2022-001438-12 (EudraCT Number)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects; Crohns Disease
Keywords: AZD7798; Single ascending dose; Repeat dose; Sentinel dosing
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Part 1a - Cohort 1: AZD7798 dose 1 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 2: AZD7798 dose 2 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 3: AZD7798 dose 3 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 4: AZD7798 dose 4 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 5: AZD7798 dose 5 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 6: AZD7798 dose 6 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Cohort 7: AZD7798 dose 7 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1b - Cohort 8: AZD7798 dose 8 (Experimental): A total of 6 subjects will receive repeat doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 1a - Spare Cohort 9: AZD7798 dose 9 (Experimental): A total of 6 subjects will receive a single ascending dose of AZD7798.
  Interventions: Biological: AZD7798
- Part 2 - Cohort 10: AZD7798 + AZD7798 (Experimental): A total of 4 subjects will receive a single dose on Day 1 followed by a single dose on Day 15.
  Interventions: Biological: AZD7798
- Part 2 - Cohort 11: Placebo + AZD7798 (Experimental): A total of 2 subjects will receive placebo on day 1 followed by AZD7798 on day 15.
  Interventions: Biological: AZD7798
- Part 2 - Cohort 12: AZD7798 + Placebo (Experimental): A total of 2 subjects will receive AZD7798 on day 1 followed by placebo on day 15.
  Interventions: Biological: AZD7798
- Placebo: Part 1a and Part 1b (Experimental): A total of 2 subjects per cohort will receive placebo.
  Interventions: Biological: Placebo
- Part 3a - Cohort 12: AZD7798 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Part 3b - Cohort 13: AZD7798 (Experimental): A total of 6 subjects will receive single ascending doses of AZD7798.
  Interventions: Biological: AZD7798
- Placebo: Part 3a and Part 3b (Experimental): A total of 2 subjects per cohort will receive placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AZD7798 — Subjects will receive AZD7798 as a single ascending dose or as a repeat dose.
  Arms: Part 1a - Cohort 1: AZD7798 dose 1; Part 1a - Cohort 2: AZD7798 dose 2; Part 1a - Cohort 3: AZD7798 dose 3; Part 1a - Cohort 4: AZD7798 dose 4; Part 1a - Cohort 5: AZD7798 dose 5; Part 1a - Cohort 6: AZD7798 dose 6; Part 1a - Cohort 7: AZD7798 dose 7; Part 1a - Spare Cohort 9: AZD7798 dose 9; Part 1b - Cohort 8: AZD7798 dose 8; Part 2 - Cohort 10: AZD7798 + AZD7798; Part 2 - Cohort 11: Placebo + AZD7798; Part 2 - Cohort 12: AZD7798 + Placebo; Part 3a - Cohort 12: AZD7798; Part 3b - Cohort 13: AZD7798
Biological: Placebo — Subjects will receive placebo matching the AZD7798 dose as a single ascending dose or as a repeat dose.
  Arms: Placebo: Part 1a and Part 1b; Placebo: Part 3a and Part 3b

SUMMARY:
This study will assess the safety, tolerability, immunogenicity, and pharmacokinetics (PK), and explore the pharmacodynamics (PD) following single ascending dose administration and repeat dose administration in healthy subjects and patients with Crohn's disease.

DETAILED DESCRIPTION:
This is a Phase I, randomised, double-blind, placebo controlled study in healthy male and female subjects as well as patients with Crohn's disease performed at a single study centre.

This study is comprised of 3 parts: Part 1 (sub-parts 1a and 1b), Part 2, and Part 3 (sub-Parts 3a and 3b).

* Part 1a: This is a First-In-Human (FIH), single ascending dose (SAD) sequential group study. Up to 7 dose levels of AZD7798 are planned to be investigated. Depending on the findings, an additional dose may be added. Up to 80 healthy subjects are planned to be included. Eight subjects will participate in each single dose cohort. Within each cohort, 6 subjects will be randomised to receive AZD7798, and 2 subjects will be randomised to receive placebo. Each subject will be enrolled up to 113 days (approximately 16 weeks).
* Part 1b: Up to 8 subjects will be randomised to receive a planned dose of AZD7798 (up to 6 subjects) or placebo (up to 2 subjects) on Day 1 and Day 15. This cohort is planned to start after completion of the single dose level cohort in Part 1a. Each subject will be enrolled up to 149 days (approximately 21 weeks).
* Part 2: Up to 8 patients will be randomised (2:1:1) into 1 of 3 strata and receive:

  * Stratum 1: AZD7798 on Day 1 and Day 15 (up to 4 patients).
  * Stratum 2: Placebo on Day 1 and AZD7798 on Day 15 (up to 2 patients).
* Stratum 3: AZD7798 on Day 1 and placebo on Day 15 (up to 2 patients). Each subject will be enrolled up to 149 days (approximately 21 weeks).
* Part 3: Subjects will be randomised to AZD7798 or placebo in a ratio of 3:1 (up to 6 subjects will receive AZD7798 and up to 2 subjects will receive placebo).

ELIGIBILITY:
Inclusion Criteria:

All Study Parts:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Subjects must have suitable veins for cannulation or repeated venepuncture.
* Males who are sexually active with a female partner of childbearing potential and who have not had a vasectomy must agree to comply with highly effective methods of contraception from the time of IMP administration until 4 months after the last dose of IMP.
* Non-smoker, or mild smoker (no more than 10 cigarettes per day).
* Have a BMI between 18 and 30 kg/m2 inclusive and weigh at least 45 kg and no more than 100 kg inclusive.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating.
* Provision of signed, written and dated informed consent for optional genetic/biomarker research.
* Evidence of completion of an appropriate vaccination regimen to SARS-CoV-2 at least 14 days prior to screening as appropriate and recommended in contemporaneous local, regional, or national guidelines.

Part 1 (Healthy Subjects), Part 3a (Healthy Japanese Subjects) and Part 3b (Healthy Chinese Subjects):

• Healthy male and female (of childbearing and non childbearing potential) subjects aged 18 to 50 years inclusive.

Part 1a (in case of dose escalation in patients) and Part 2 (Patients with Crohn's Disease):

* Male and female (of childbearing and non childbearing potential) patients with Crohn's disease aged 18 to 60 years inclusive.
* Patients with confirmed Crohn's disease (diagnosed via endoscopy, histology and/or imaging) with onset of symptoms at least 3 months prior to screening.
* Active disease, defined by at least one symptom and sign consistent with Crohn's disease AND at least one of the following:

  1. CRP > 5mg/L at screening.
  2. Faecal calprotectin > 250μg/g at screening.
  3. Evidence of active inflammation on cross-sectional imaging within past 3 months prior to screening.
  4. Evidence of active inflammation on endoscopy within past 3 months prior to screening.

Part 3a (Japanese Subjects) • Subject is a native of Japan; defined as having both parents and 4 grandparents who are Japanese. This includes second and third generation subjects of Japanese descent whose parents or grandparents are living in a country other than Japan.

Part 3b (Chinese Subjects)

* Healthy Chinese subjects. Subjects of Chinese ancestry are eligible based on meeting all of the following:

  1. Born in mainland China, Hong Kong, or Taiwan.
  2. Descendants of 4 ethnic Chinese grandparents and 2 ethnic Chinese parents.
  3. Have lived outside China for less than 10 years at the time of screening.

     Exclusion Criteria:

     All Study Parts:

     • Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational Medicinal Product (IMP).

     • Any positive result on Screening for HBsAg, anti-HBc antibody, anti-HCV antibody, and HIV.

     • History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or, history of hypersensitivity to drugs with a similar chemical structure or class to AZD7798.

     • For females of childbearing potential using hormonal contraception: Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.

     • Subjects with a positive diagnostic nucleic acid test (using PCR) for SARS-CoV-2 prior to dosing.

     • Live or attenuated vaccine within 4 weeks of Visit 1 and until the end of the follow up period.
     * An active infection, or history of serious infection within the preceding 28 days.
     * Use of antibiotics within 28 days prior to the first administration of IMP.
     * History of symptomatic herpes simplex (excluding cold sores) or herpes zoster infection within 3 months prior to screening.
     * Positive or indeterminate TB QuantiFERON test.
     * Has received another new chemical entity within 30 days/5 half-lives of the first administration of IMP in this study.
     * Subjects who cannot communicate reliably with the Investigator.
     * Vulnerable subjects.

     Part 1 (Healthy Subjects), Part 3a (Japanese Subjects, and Part 3b (Chinese Subjects):

     • Any laboratory values with deviations.

     • Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results other than those described under exclusion criterion number 20, as judged by the Investigator.

     • Abnormal vital signs, after 5 minutes supine rest at screening and admission.

     • Known or suspected history of drug abuse in the last 1 year as judged by the Investigator.

     • History of alcohol abuse or excessive intake of alcohol within the last 1 year. as judged by the Investigator.

     • Positive screen for drugs of abuse at screening or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit prior to the first administration of the IMP.

     • Excessive intake of caffeine containing drinks or food (eg, coffee, tea, chocolate,) as judged by the Investigator.

     Part 1a (in case of dose escalation in patients) and Part 2 (Patients with Crohn's Disease):

     • Patients with any uncontrolled medical conditions, other than active Crohn's disease, that in the opinion of the Investigator put the patient at unacceptable risk or interfere with study assessments or integrity of the data.

     • Current diagnosis of ulcerative colitis, indeterminate colitis, inflammatory bowel disease-unclassified, infectious colitis, or ischaemic colitis.

     • History of CMV colitis 12 months prior to screening.

     • Patients with fulminant Crohn's disease or toxic megacolon.

     • Planned surgery for Crohn's disease prior to the end of study follow up visit.

     • Patients with symptomatic intestinal stenosis, known pre-stenotic dilatation, undrained fistula(e), or abscesses.

     • Initiation or change in dose of azathioprine or mercaptopurine (including initiation or discontinuation of allopurinol) within 4 weeks of the first administration of IMP.

     • Treatment with methotrexate, ciclosporin, tacrolimus or thalidomide within 4 weeks of the first administration of IMP.

     • Treatment with an anti-TNF biologic within 8 weeks of the first administration of IMP, unless therapeutic drug monitoring is performed and drug concentrations are undetectable.
     * Treatment with any biologic, other than an anti-TNF, within 12 weeks or with undetectable serum concentrations prior to the first administration of IMP, unless therapeutic drug monitoring is performed and drug concentrations are undetectable.
     * Treatment with rituximab within 12 months prior to the first administration of IMP.
     * Any laboratory values with deviations.
     * Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results other than those described under exclusion criterion number 49, as judged by the Investigator.
     * Abnormal vital signs, after 5 minutes supine rest, defined as any of the following at screening and admission.
     * Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12 lead ECG.
     * Unstable lifestyle factors, such as alcohol use to excess or recreational drug use, to the extent that in the opinion of the Investigator they would interfere with the ability of a patient to complete the study.
     * Current malignancy or history of malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Until follow-up (Day 85) or Early termination (ET)
  The safety and tolerability of AZD7798 following administration of single ascending doses will be assessed.

SECONDARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The AUCinf of AZD7798 following administration of single ascending doses will be assessed.
AUClast | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The AUClast of AZD7798 following administration of single ascending doses will be assessed.
Maximum serum concentration (Cmax) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The Cmax of AZD7798 following administration of single ascending doses will be assessed.
Time to reach maximum serum concentration (tmax) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The tmax of AZD7798 following administration of single ascending doses will be assessed.
Time to last measurable concentration (tlast) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The tlast of AZD7798 following administration of single ascending doses will be assessed.
Terminal elimination half-life (t½λz) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The t½λz of AZD7798 following administration of single ascending doses will be assessed.
Systemic clearance (CL) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The CL of AZD7798 following administration of single ascending doses will be assessed.
Apparent total clearance (CL/F) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The CL/F of AZD7798 following administration of single ascending doses will be assessed.
Volume of distribution based on the terminal phase (Vz) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The Vz of AZD7798 following administration of single ascending doses will be assessed.
Apparent volume of distribution based on terminal phase (Vz/F) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The Vz/F of AZD7798 following administration of single ascending doses will be assessed.
Bioavailability (F) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The F of AZD7798 following administration of single ascending doses will be assessed.
Volume of distribution at steady state (Vss) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The Vss of AZD7798 following administration of single ascending doses will be assessed.
AUClast/D | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The AUClast/D of AZD7798 following administration of single ascending doses will be assessed.
AUCinf/D | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The AUCinf/D of AZD7798 following administration of single ascending doses will be assessed.
Cmax/D | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The Cmax/D of AZD7798 following administration of single ascending doses will be assessed.
Percentage of patients with antidrug antibodies (ADAs) | Day 1 to Day 8, and Days 15, 22, 29, 43, 57, and 85
  The immunogenicity of AZD7798 following administration of single ascending doses will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D9690C00001_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9690C00001&attachmentIdentifier=5a1bca35-fbcf-4b96-a545-f21225c41efd&fileName=D9690C00001_CSR_synopsis_Redacted.pdf&versionIdentifier=